CLINICAL TRIAL: NCT06437379
Title: Effect of Teaching Protocol on Nurse's Knowledge and Practice Regarding Infection Control Measures for Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Infection Control Measures for Patients Undergoing Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kamilia Farouk Abdel Fattah Osman, Nursing specialist, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Infection Control Measures
Record Dates: First submitted 2024-03-17; First posted 2024-05-31 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2024-03

CONDITIONS: Urological Nursing; Kidney Stone
Keywords: PCNL; infection control; nurses
MeSH Terms: conditions — Kidney Calculi | interventions — Infection Control

STUDY DESIGN:
Intervention Model Description: To evaluate the effect of implementing teaching protocol on nurse's knowledge and practice regarding infection control measures for patients undergoing Percutaneous Nephrolithotomy.
Masking Description: nurse working in urology department
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- effect of infection control on patient outcomes undergoing PCNL (Experimental): Effect of Teaching Protocol on Nurse's Knowledge and Practice regarding Infection Control Measures for Patients undergoing Percutaneous Nephrolithotomy
  Interventions: Behavioral: Infection control

INTERVENTIONS:
Behavioral: Infection control — To evaluate the effect of implementing teaching protocol on nurse's knowledge and practice regarding infection control measures for patients undergoing Percutaneous Nephrolithotomy.

SUMMARY:
To evaluate the effect of implementing teaching protocol on nurse's knowledge and practice regarding infection control measures for patients undergoing Percutaneous Nephrolithotomy.

DETAILED DESCRIPTION:
Percutaneous Nephrolithotomy (PCNL) is a surgery to remove kidney stones that are too large to pass on their own. Percutaneous" means that the procedure occurs through the skin. "Nephrolithotomy" means the removal of a calculus (kidney stone) from a kidney . Percutaneous Nephrolithotomy is typically recommended when kidney stones are larger than 0.8 inch (2 centimeters) in diameter. . Percutaneous Nephrolithotomy (PCNL) has altered dramatically the management of urolithiasis. In fact, these treatment modalities have nearly 99% success rates for treatment of upper urinary tract stones. . There were several complications related to Percutaneous Nephrolithotomy such as fever (23%) and bleeding necessitating transfusion (12%). Extravasation was seen in 7% of patients and transient ureteral obstruction in 6%. The complications limit surgical outcome of PCNL. Infection remains the most common complication arising from this procedure and some patients develop septicemia and septic shock, resulting in increased mortality and morbidity. So, the success of the Percutaneous Nephrolithotomy depends on the maintenance of infection control precautions. This is why investigator looked at this study. Knowledge of the nurse of percutaneous nephrolithotomy care was of crucial importance and had an impact on nurse's practice. The main goal of care was to prevent infection undergoing the percutaneous nephrolithotomy The nurses' role preventing infection for patient undergoing (PCNL) and mainly maintain the sterile field and after operation safety removing (PPE), washing instruments used during operation all of that resulting in positive surgical outcomes Infection control is an important concern for health care professionals specially nurses. Nurses have higher risk for both self-acquiring and transmitting infections to other patients infection control practices form the backbone of nurse's. Nurses has the distinctive opportunity to reduce hospital - acquired infections by utilizing the skills and knowledge about infection control measures, they can facilitate patient recovery while minimizing complications related to infections. Compliance with infection control and sterile technique principles will be prevent nosocomial infections in the operating room, and the patient's hospital stay being shorter and a reduced cost for the medical aids and hospitals . the investigators searched for this topic in many sites such as PubMed Central, Research Gate, and Science.gov.The current topic was not covered in the previous studies. Previous studies did not include specific point about this topic but include general point about PCNL and this strong rational for this study. This study will be carried out to evaluate the knowledge and practice about standard precautions and infection control measures and to explore education needs of nurses.

Generally, programs of healthcare education vary greatly in their contents and approaches .Various forms of visual aids are currently used in healthcare education including illustrations such as photographs and animations such as computer -generated clips and video clips.

ELIGIBILITY:
Inclusion Criteria:

1- Nursing Staff providing nursing care services for patient undergoing PNL (pre-intra-post) operative care.

Exclusion Criteria:

1. Head nurses
2. Nurses refused to participate in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
teach nurses new measures to reduce infection in patient undergoing PCNL by applying infection control measure | one year
  use infection control technique to reduce infection in patient undergoing PCNL

SECONDARY OUTCOMES:
reduce the patients hospital stay postoperative | one year
  reduce patient length of hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babjuk M, Burger M, Capoun O, Cohen D, Comperat EM, Dominguez Escrig JL, Gontero P, Liedberg F, Masson-Lecomte A, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Seisen T, Soukup V, Sylvester RJ. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (Ta, T1, and Carcinoma in Situ). Eur Urol. 2022 Jan;81(1):75-94. doi: 10.1016/j.eururo.2021.08.010. Epub 2021 Sep 10. PMID 34511303